CLINICAL TRIAL: NCT02546921
Title: A Cancer Research UK Phase I Study of MOv18 IgE, a First in Class Chimeric IgE Antibody Against Folate Receptor-alpha, in Patients With Advanced Solid Tumours
Brief Title: Phase I Study of MOv18 IgE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRUKD/14/001; 2014-000070-19 (EudraCT Number)
Record Dates: First submitted 2015-08-19; First posted 2015-09-11 (Estimated); Results first posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2022-07

CONDITIONS: Human Cancers
Keywords: IgE antibody; Folate receptor; Cancer Immunotherapy; First in class

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- MOv18 IgE Cohort 1 (Experimental)
  Interventions: Drug: MOv18 IgE
- MOv18 IgE Cohort 2 (Experimental)
  Interventions: Drug: MOv18 IgE
- MOv18 IgE Cohort 3 (Experimental)
  Interventions: Drug: MOv18 IgE
- MOv18 IgE Cohort 4 (Experimental)
  Interventions: Drug: MOv18 IgE
- MOv18 IgE Cohort 5 (Experimental)
  Interventions: Drug: MOv18 IgE
- MOv18 IgE Cohort 6 (Experimental)
  Interventions: Drug: MOv18 IgE
- MOv18 IgE Cohort 7 (Experimental)
  Interventions: Drug: MOv18 IgE

INTERVENTIONS:
Drug: MOv18 IgE — The allocated dose of 70 µg MOv18 IgE will be diluted in 250 mL saline and administered by IV infusion once weekly for 6 weeks, followed by fortnightly for 6 weeks if the patient appears to be benefiting from MOv18 IgE. Each IV infusion will be preceded by an intradermal injection of 0.1 mL of a 2 µg/mL MOv18 IgE solution for safety assessment.
  Arms: MOv18 IgE Cohort 1
Drug: MOv18 IgE — The allocated dose of 250 µg MOv18 IgE will be diluted in 250 mL saline and administered by IV infusion once weekly for 6 weeks, followed by fortnightly for 6 weeks if the patient appears to be benefiting from MOv18 IgE. Each IV infusion will be preceded by either an intradermal injection of 0.1 mL of a 2 µg/mL MOv18 IgE solution or a skin prick test with 2 µg/mL MOv18 IgE solution, for safety assessment.
  Arms: MOv18 IgE Cohort 2
Drug: MOv18 IgE — The allocated dose of 500 µg MOv18 IgE will be diluted in 250 mL saline and administered by IV infusion once weekly for 6 weeks, followed by fortnightly for 6 weeks if the patient appears to be benefiting from MOv18 IgE. Each IV infusion will be preceded by a skin prick test with 2 µg/mL MOv18 IgE solution, for safety assessment.
  Arms: MOv18 IgE Cohort 3
Drug: MOv18 IgE — The allocated dose of 700 µg MOv18 IgE will be diluted in 250 mL saline and administered by IV infusion once weekly for 6 weeks, followed by fortnightly for 6 weeks if the patient appears to be benefiting from MOv18 IgE. Each IV infusion will be preceded by a skin prick test with 2 µg/mL MOv18 IgE solution, for safety assessment.
  Arms: MOv18 IgE Cohort 4
Drug: MOv18 IgE — The allocated dose of 1.5 mg MOv18 IgE will be diluted in 250 mL saline and administered by IV infusion once weekly for 6 weeks, followed by fortnightly for 6 weeks if the patient appears to be benefiting from MOv18 IgE. Each IV infusion will be preceded by a skin prick test with 2 µg/mL MOv18 IgE solution, for safety assessment.
  Arms: MOv18 IgE Cohort 5
Drug: MOv18 IgE — The allocated dose of 3 mg MOv18 IgE will be diluted in 250 mL saline and administered by IV infusion once weekly for 6 weeks, followed by fortnightly for 6 weeks if the patient appears to be benefiting from MOv18 IgE. Each IV infusion will be preceded by a skin prick test with 2 µg/mL MOv18 IgE solution, for safety assessment.
  Arms: MOv18 IgE Cohort 6
Drug: MOv18 IgE — Cycle 1 - The allocated dose of 6 mg MOv18 IgE will be diluted in 250 mL saline and administered by IV infusion once weekly for 3 weeks.
  Cycle 2 - The allocated dose of 12 mg MOv18 IgE will be diluted in 250 mL saline and administered by IV infusion once weekly for 3 weeks, followed by fortnightly for 6 weeks if the patient appears to be benefiting from MOv18 IgE.
  Each IV infusion will be preceded by a skin prick test with 2 µg/mL MOv18 IgE solution, for safety assessment.
  Arms: MOv18 IgE Cohort 7

SUMMARY:
This first in human study of the new therapeutic antibody MOv18 immunoglobulin (Ig) E, which targets a protein called folate receptor alpha (FRa), in patients with advanced cancer seeks to demonstrate the potential for the use of this IgE antibody as an example of the use of the IgE class of antibodies for the treatment of cancer.

DETAILED DESCRIPTION:
Therapeutic antibodies have significantly improved the prognosis of patients with a range of cancers. Currently available therapeutic antibodies belong to the IgG class. This study is looking at a new drug called MOv18 IgE which belongs to a different class of antibody, the IgE class. IgE antibodies may trigger a more powerful immune response to tumour cells than these available IgG antibodies and so be more effective in treating certain types of cancer. This is the first time an IgE antibody therapy will be given to patients with cancer.

The MOv18 IgE antibody is designed to recognise and attach to FRa. Scientists have found more of this protein on the surface of certain cancer cells than on the surface of normal cells, most commonly ovarian cancer but also cancers of the kidney, endometrium, lung, breast, bladder, colon and pancreas. Once attached, the MOv18 IgE antibody should trigger the body's own immune system to attack and kill the cancer cells.

Patients will be selected based on the presence of FRa on their tumour in a previous biopsy. The study is the first study of this new antibody treatment to be given to humans and will focus primarily on the assessment of safety confirming the findings of preclinical studies that exposure to MOv18 IgE will not trigger anaphylaxis. This is in addition to extensive pharmacokinetic (PK), biodistribution of the antibody and immunological response. The study will follow a dose escalation design where small groups of patients are treated at a set dose, starting with a very low dose followed by exponential increasing doses, to find a safe dose at which the drug has a good chance of effectively treating the cancer. Patients will receive a short course of treatment. Patients treated at the higher dose levels will be asked to provide a pre and post treatment biopsy to explore the effect of the treatment on the tumour.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically-proven advanced, unresectable solid tumour of a type known to express FRα in a percentage of cases
2. Archival tumour tissue expressing FRα (1+, 2+ or 3+ membrane staining on at least 5% of tumour cells by immunohistochemistry using the BN3.2 antibody, based on the technique described by Lawson & Scorer, 2010).
3. Advanced disease for which no alternative therapy is felt to be appropriate.
4. Measurable disease or disease evaluable by tumour marker. Measurable disease is preferred for patients entering higher cohorts to facilitate efficacy assessments.
5. World Health Organisation (WHO) performance status of 0 or 1 and a life expectancy of at least 12 weeks.
6. Haematological and biochemical indices within the ranges shown below. These measurements should be performed within 7 days before the first dose of MOv18 IgE (Day -7 to Pre-dose on Day 1). Measurements performed before Day -7 may be accepted by the CDD to demonstrate eligibility if repeat testing is logistically difficult for the patient and is not considered necessary medically in the opinion of the Investigator or CDD.

   Laboratory Test Value required Haemoglobin (Hb) ≥ 9.0 g/dL Absolute neutrophil count ≥ 1.5 x 10^9/L Platelet count ≥ 100 x 10^9/L Serum bilirubin ≤ 1.5 x upper limit of normal (ULN) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN unless raised due to liver metastases in which case up to 5 x ULN is permissible Serum creatinine ≤ 1.5 x ULN
7. Aged 16 years or over at the time consent is given.
8. Written (signed and dated) informed consent and capable of co-operating with treatment and follow-up.

Exclusion Criteria:

1. Radiotherapy (except for palliative reasons), endocrine therapy, immunotherapy or chemotherapy during the previous four weeks (six weeks for nitrosoureas and mitomycin-C) and investigational medicinal products during the previous 4 weeks, or 5 product half-lives before treatment.
2. Patients on beta-blockers and unable to interrupt beta-blockade (which may counteract the therapeutic effects of adrenaline), or tricyclic anti-depressants/MAOIs (which can dangerously augment the effects of adrenaline). These agents should be discontinued at least 4 half-lives before administration of the first dose of MOv18 IgE and for the duration of MOv18 IgE therapy.
3. Patients on bisphosphonates or treated with bisphosphonates in the last 18 months.
4. Ongoing toxic manifestations of previous treatments that have not resolved to Grade 1 or lower (other than alopecia of any grade or Grade 2 peripheral neuropathy).
5. Known brain metastases that have not been previously treated and been stable for at least 2 months.
6. Female patients who are able to become pregnant (or already pregnant or lactating). However, those female patients who have a negative serum or urine pregnancy test before enrolment and agree to use two highly effective forms of contraception (oral, injected or implanted hormonal contraception and condom; have an intra-uterine device and condom; diaphragm with spermicidal gel and condom) effective at the first administration of IMP, throughout the study and for six months afterwards are considered eligible.
7. Male patients with partners of child-bearing potential (unless they agree to take measures not to father children by using one form of highly effective contraception at the first administration of IMP, throughout the study and for six months afterwards) or agree to sexual abstinence*. Men with pregnant or lactating partners should be advised to use barrier method contraception (for example, condom plus spermicidal gel) to prevent exposure to the foetus or neonate.

   * Abstinence is only considered to be an acceptable method of contraception when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
8. Major thoracic or abdominal surgery from which the patient has not yet recovered.
9. At high risk from the effects of anaphylaxis because of non-malignant systemic disease including active uncontrolled infection, cardiac failure, peripheral vascular disease, previous cerebrovascular accident (CVA), dyspnoea due to heart failure, extensive lung metastases, significant pleural effusions or other conditions.
10. History of laryngeal oedema, uncontrolled or high risk asthma (according to Global Initiative for Asthma (GINA) guidelines), or anaphylaxis. Patients with a history of hypersensitivity to carboplatin, taxanes, or contrast media may enter the study at the investigator's discretion.
11. Patients with any congenital or acquired immunodeficiency syndrome or receiving immunosuppressive therapy (including any dose of systemic corticosteroids), or who are immunosuppressed post organ transplant. However, patients receiving inhaled corticosteroids and patients with a history of allergy (other than anaphylaxis) are eligible, as are patients with a history of auto-immune disease.
12. Known to be serologically positive for hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
13. Patients with baseline elevation in serum tryptase (indicating possible mastocytosis) or a positive baseline basophil activation test (indicating a hypothetical potential for anaphylaxis with MOv18 IgE).
14. Participating or planning to participate in another interventional clinical trial, whilst taking part in this study. Participation in an observational study or in the follow-up phase of a previous interventional trial is acceptable.
15. Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical study.
16. Patients unwilling or unable to interrupt antihistamines (which may interfere with skin prick testing). Antihistamines should be discontinued at least 4 half-lives before the first skin prick test.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Spicer, Dr, Principal Investigator — Guy's and St Thomas's Hospital
Locations (4):
- United Kingdom (4):
  - Addenbrooke's Hospital, Cambridge, Cambridge
  - Guy's and St Thomas's Hospital, London
  - University College London Hospital, London
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stavraka C, Chauhan J, Crescioli S, McSweeney SM, Pope A, Gillett C, Di Meo A, Prassas I, Laddach R, Stoker K, McCraw AJ, Adams R, Tull TJ, Naban N, Willsmore Z, Semkova KV, Grattan CEH, McGrath J, Till SJ, Corrigan CJ, Kristeleit R, Tsoka S, Diamandis EP, Lacy KE, Pinder S, Josephs DH, Spicer J, Bax HJ, Karagiannis SN. Non-Allergic Urticarial Skin Reactions Associated With MOv18 IgE, a First-In-Class IgE Antibody Recognising Folate Receptor Alpha. Allergy. 2025 Aug;80(8):2225-2239. doi: 10.1111/all.16514. Epub 2025 Mar 6. PMID 40045925
- [Derived] Spicer J, Basu B, Montes A, Banerji U, Kristeleit R, Miller R, Veal GJ, Corrigan CJ, Till SJ, Figini M, Canevari S, Barton C, Jones P, Mellor S, Carroll S, Selkirk C, Nintos G, Kwatra V, Funingana IG, Doherty G, Gould HJ, Pellizzari G, Nakamura M, Ilieva KM, Khiabany A, Stavraka C, Chauhan J, Gillett C, Pinder S, Bax HJ, Josephs DH, Karagiannis SN. Safety and anti-tumour activity of the IgE antibody MOv18 in patients with advanced solid tumours expressing folate receptor-alpha: a phase I trial. Nat Commun. 2023 Jul 25;14(1):4180. doi: 10.1038/s41467-023-39679-9. PMID 37491373
- See also: Simple summary of trial on Cancer Research UK Trial Database — http://www.cancerresearchuk.org/about-cancer/find-a-clinical-trial/a-trial-looking-at-mov18-ige-for-advanced-solid-tumours
- See also: Interim phase 1 data evaluating MOv18 IgE, an anti-folate receptor alpha IgE antibody, in cancer patients with advanced solid tumours presented at the AACR Virtual Annual Meeting I — http://www.alsaventures.com/news/epsilogen-press-release

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial participants were enrolled at four trial sites between 18 November 2015 and 05 August 2021.
Period: Overall Study
Arm/Group | MOv18 IgE Cohort 1 | MOv18 IgE Cohort 2 | MOv18 IgE Cohort 3 | MOv18 IgE Cohort 4 | MOv18 IgE Cohort 5 | MOv18 IgE Cohort 6 | MOv18 IgE Cohort 7
Started | 2 | 8 | 6 | 3 | 3 | 3 | 1
Completed | 1 | 2 | 4 | 3 | 2 | 2 | 1
Not Completed | 1 | 6 | 2 | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 5 | 2 | 0 | 0 | 0 | 0
Not completed — Evidence of Disease Progression | 1 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Patient Choice | 0 | 1 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MOv18 IgE Cohort 1 | MOv18 IgE Cohort 2 | MOv18 IgE Cohort 3 | MOv18 IgE Cohort 4 | MOv18 IgE Cohort 5 | MOv18 IgE Cohort 6 | MOv18 IgE Cohort 7 | Total
Number analyzed (Participants) | 2 | 8 | 6 | 3 | 3 | 3 | 1 | 26
Age, Continuous [Median (Full Range); unit: years] | 61 [52 to 70] | 58.5 [47 to 66] | 59.5 [53 to 71] | 65 [64 to 79] | 54 [51 to 58] | 63 [55 to 69] | 75 [75 to 75] | 60 [47 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 8 | 6 | 3 | 3 | 3 | 1 | 26
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 2 | 8 | 6 | 3 | 3 | 3 | 1 | 26

OUTCOME MEASURES:

1. Primary Outcome: Serious Adverse Events (SAEs) and Non-serious Adverse Events (AEs) Considered to be at Least Possibly Related to MOv18 IgE
Description: Reported safety information in the form of AEs, categorised according to Medical Dictionary for Regulatory Activities (MedDRA) version (v) 24.0 and graded for severity according to National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.02. AEs will be assessed by the reporting study doctors for a causal relationship to MOv18 IgE. Count of AEs by arm.
Time Frame: From the date of written informed consent and until the end of safety follow up period for MOv18 IgE, a median of 88.5 days (range: 13 to 181 days).
Population: All enrolled participants who received at least one dose of MOv18 IgE by IV infusion, intradermally or as a skin prick test.
Measure: Count of Participants; unit: Participants
Arm/Group | MOv18 IgE Cohort 1 | MOv18 IgE Cohort 2 | MOv18 IgE Cohort 3 | MOv18 IgE Cohort 4 | MOv18 IgE Cohort 5 | MOv18 IgE Cohort 6 | MOv18 IgE Cohort 7
Number analyzed (Participants) | 2 | 8 | 6 | 3 | 3 | 3 | 1
Participants
  No. participants at least one Related SAEs | 0 | 5 | 2 | 0 | 0 | 1 | 0
  No. participants at least one Related NSAEs | 0 | 5 | 5 | 3 | 3 | 3 | 1

2. Primary Outcome: Number of Participants Who Experienced Dose Limiting Toxicities (DLTs)
Description: DLTs graded for severity using the NCI CTCAE v4.02, measured by count of participants per arm. Two DLTs were reported; however, following review of the data, it was determined that events of this nature did not constitute DLTs. The trial protocol was updated so that if further similar events occurred then would not be considered as DLTs but the events already reported remain categorised as DLTs.
Time Frame: From first dose onwards until completion of Cycle 1 (3 weeks).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MOv18 IgE Cohort 1 | MOv18 IgE Cohort 2 | MOv18 IgE Cohort 3 | MOv18 IgE Cohort 4 | MOv18 IgE Cohort 5 | MOv18 IgE Cohort 6 | MOv18 IgE Cohort 7
Number analyzed (Participants) | 2 | 8 | 6 | 3 | 3 | 3 | 1
Participants | 0 | 1 | 1 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Dose Independent Significant Toxicities
Description: AEs judged to be due to systemic mast cell degranulation (i.e. anaphylaxis). No dose independent significant toxicities were reported. However, one event of anaphylactic reaction was classified as a DLT at the time of occurrence but, following review of the data, the trial protocol was updated. This meant that any future events of anaphylaxis would have been classified as dose independent toxicities, but the event already reported remained as a DLT.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Dose Independent Significant Toxicities
Arm/Group | MOv18 IgE Cohort 1 | MOv18 IgE Cohort 2 | MOv18 IgE Cohort 3 | MOv18 IgE Cohort 4 | MOv18 IgE Cohort 5 | MOv18 IgE Cohort 6 | MOv18 IgE Cohort 7
Number analyzed (Participants) | 2 | 8 | 6 | 3 | 3 | 3 | 1
Dose Independent Significant Toxicities | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Grade ≥2 Laboratory Parameter AEs Reported
Description: Reported safety information in the form of haematological or biochemical abnormalities that were reported as AEs and graded for severity according to NCI CTCAE v4.02.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MOv18 IgE Cohort 1 | MOv18 IgE Cohort 2 | MOv18 IgE Cohort 3 | MOv18 IgE Cohort 4 | MOv18 IgE Cohort 5 | MOv18 IgE Cohort 6 | MOv18 IgE Cohort 7
Number analyzed (Participants) | 2 | 8 | 6 | 3 | 3 | 3 | 1
Participants
  No. participants at least one Biochem Grade >=2 AE | 0 | 0 | 1 | 0 | 0 | 0 | 0
  No. participants at least one Haem Grade >=2 AE | 0 | 4 | 2 | 0 | 0 | 0 | 0

5. Secondary Outcome: Antitumour Activity (Best Response) of MOv18 IgE Measured According to the Response Evaluation Criteria in Solid Tumours (RECIST) v 1.1
Description: Best radiological response observed according to RECIST v1.1, presented per arm by count of participants. RECIST responses include complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD). For a response to be defined as SD, the criteria must have been met at least once at a minimum interval of 6 weeks after study entry.
Time Frame: Radiological disease response assessment at screening/baseline and every 6 weeks to end of treatment, a median of 56.5 days (range: 38 to 124 days).
Population: Eligible participants who received at least one complete IV dose of MOv18 IgE and had a baseline and at least one post-baseline assessment of disease according to RECIST v1.1. Although 13 participants were initially reported to have a best response of SD, 2 of these participants were not evaluable for SD, as the assessment was performed <6 weeks after the first IV infusion of MOv18 IgE. Therefore, the total number (%) of participants with SD is reported here as 11 (55.0%).
Measure: Count of Participants; unit: Participants
Groups:
- MOv18 IgE Cohorts 1 - 7: The allocated dose of MOv18 IgE (70μg-12mg) will be diluted in 250 mL saline and administered by IV infusion once weekly for three weeks (6 mg and 12 mg) or six weeks (70 μg-3 mg), followed by fortnightly for six weeks (all dose levels except 6mg) if the patient appears to be benefiting from MOv18 IgE. Each IV infusion will be preceded by either an intradermal injection of 0.1 mL of a 2 μg/mL MOv18 IgE solution or a skin prick test with 2 μg/mL MOv18 IgE solution, for safety assessment.
Arm/Group | MOv18 IgE Cohorts 1 - 7
Number analyzed (Participants) | 26
Participants
  Stable disease | 11
  Progressive disease | 7
  Not evaluable | 2

6. Secondary Outcome: Antitumour Activity Measured by the Percentage Change in Cancer Antigen 125 (CA125) Tumour Marker Levels During the Trial, in Participants With Elevated CA125 at Baseline
Description: The percentage change in CA125 levels from baseline to the last measurement taken on-treatment, presented as a median (minimum, maximum) for each arm.
Time Frame: Disease response assessment at screening/baseline and every six weeks, if clinically appropriate for tumour type, to end of treatment, for a median of 34 days (range: 5 to 91 days).
Population: All eligible participants who received at least one complete IV dose of MOv18 IgE and who had elevated CA125 at baseline (>35 kU/L).
Measure: Median (Full Range); unit: % change from baseline CA125 level
Arm/Group | MOv18 IgE Cohort 1 | MOv18 IgE Cohort 2 | MOv18 IgE Cohort 3 | MOv18 IgE Cohort 4 | MOv18 IgE Cohort 5 | MOv18 IgE Cohort 6 | MOv18 IgE Cohort 7
Number analyzed (Participants) | 1 | 3 | 4 | 3 | 3 | 3 | 1
% change from baseline CA125 level | 41.38 [41.38 to 41.38] | 59.04 [-14.13 to 227.52] | 52.79 [15.12 to 80.36] | 118.13 [-32.31 to 264.9] | 45.41 [14.75 to 100.41] | 15.93 [13.82 to 31.86] | 144.14 [144.14 to 144.14]

7. Secondary Outcome: Measurement of Pharmacokinetic (PK) Parameter Area Under the Concentration-Time Curve From Time 0 to 24 Hours of MOv18 IgE
Description: Area under the serum concentration-time curve from time 0 to 24 hours after IV MOv18 IgE administration, evaluated using an enzyme linked immunosorbent assay (ELISA) method. Not all participants were analysed at all time points.
Time Frame: Cohorts 1-7: Cycle 1 Day 1 within 24 hours (h) predose, then 30 mins postdose and 2, 4, 6 and 24 h postdose. Cohort 7 only (intrapatient dose escalation): Cycle 2 Day 1 predose, then 30 mins postdose and 2, 4, 6 and 24 h postdose. Each cycle = 21 days.
Population: All participants who received a complete IV infusion of MOv18 IgE on Cycle 1, Day 1 and, for Cohort 7 only, Cycle 2 Day 1. For this outcome measure, data for Cohort 7 are reportedly separately by dose level.
Measure: Mean (Standard Deviation); unit: ng/mL.h
Groups:
- MOv18 IgE Cohort 7 Before Intra-Patient Dose Escalation: MOv18 IgE: Cycle 1 - The allocated dose of 6 mg MOv18 IgE will be diluted in 250 mL saline and administered by IV infusion once weekly for 3 weeks. If the dose is tolerated then it will be escalated for Cycle 2.
  Each IV infusion will be preceded by a skin prick test with 2 µg/mL MOv18 IgE solution, for safety assessment.
- MOv18 IgE Cohort 7 After Intra-patient Dose Escalation: MOv18 IgE: after receiving three IV infusions of 6 mg MOv18 IgE in Cycle 1, the dose will be escalated. The allocated dose of 12 mg MOv18 IgE will be diluted in 250 mL saline and administered by IV infusion once weekly for 3 weeks followed by fortnightly for 6 weeks if the patient appears to be benefiting from MOv18 IgE. Each IV infusion will be preceded by a skin prick test with with 2 μg/mL MOv18 IgE solution, for safety assessment.
Arm/Group | MOv18 IgE Cohort 1 | MOv18 IgE Cohort 2 | MOv18 IgE Cohort 3 | MOv18 IgE Cohort 4 | MOv18 IgE Cohort 5 | MOv18 IgE Cohort 6 | MOv18 IgE Cohort 7 Before Intra-Patient Dose Escalation | MOv18 IgE Cohort 7 After Intra-patient Dose Escalation
Number analyzed (Participants) | 2 | 5 | 5 | 2 | 2 | 1 | 1 | 1
ng/mL.h | NA (NA) — In one participant, MOv18 IgE could not be quantified in samples at any time point. In the other participant, MOv18 IgE could only be detected up to 7 hours postdose | 130 (76) | 303 (159) | 222 (42) | 726 (113) | 761 (NA) — Only one patient had evaluable data at this timepoint | 2134 (NA) — Only one patient had evaluable data at this timepoint | 5573 (NA) — Only one patient had evaluable data at this timepoint

8. Secondary Outcome: Measurement of PK Parameter Maximum Observed Serum Concentration (Cmax) of MOv18 IgE
Description: Cmax in serum following IV MOv18 IgE administration was analysed using an ELISA method. Not all participants were analysed at all time points.
Time Frame: Cohorts 1-7: Cycle 1 Day 1 <24 h predose, then 30 mins postdose and 2, 4, 6, 24 and 48 h postdose; Cycle 1 Day 8 predose. Cohort 7 only (intrapatient escalation): Cycle 2 Day 1 predose, then 30 mins and 2, 4, 6 and 24 h postdose. Each cycle = 21 days.
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MOv18 IgE Cohort 1 | MOv18 IgE Cohort 2 | MOv18 IgE Cohort 3 | MOv18 IgE Cohort 4 | MOv18 IgE Cohort 5 | MOv18 IgE Cohort 6 | MOv18 IgE Cohort 7 Before Intra-Patient Dose Escalation | MOv18 IgE Cohort 7 After Intra-patient Dose Escalation
Number analyzed (Participants) | 2 | 5 | 5 | 2 | 2 | 1 | 1 | 1
ng/mL | 2.3 (NA) — Only one patient had evaluable data at this timepoint | 9.4 (6.8) | 31.8 (11.4) | 29.7 (4.6) | 86.8 (18.3) | 75.7 (NA) — Only one patient had evaluable data at this timepoint | 196.7 (NA) — Only one patient had evaluable data at this timepoint | 368.2 (NA) — Only one patient had evaluable data at this timepoint

9. Secondary Outcome: Measurement of PK Parameter Time to Reach Maximum Observed Serum Concentration (Tmax) of MOv18 IgE
Description: Serum samples were analysed to determine the Tmax of MOv18 IgE following IV administration using an ELISA method. Not all participants were analysed at all time points.
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Median (Standard Deviation); unit: Hour
Arm/Group | MOv18 IgE Cohort 1 | MOv18 IgE Cohort 2 | MOv18 IgE Cohort 3 | MOv18 IgE Cohort 4 | MOv18 IgE Cohort 5 | MOv18 IgE Cohort 6 | MOv18 IgE Cohort 7 Before Intra-Patient Dose Escalation | MOv18 IgE Cohort 7 After Intra-patient Dose Escalation
Number analyzed (Participants) | 2 | 5 | 5 | 2 | 2 | 1 | 1 | 1
Hour | 3.5 (NA) — Only one patient had evaluable data at this timepoint | 2.2 (0.6) | 2.2 (0.5) | 2.2 (0.1) | 2.0 (0.3) | 2.1 (NA) — Only one patient had evaluable data at this timepoint | 1.0 (NA) — Only one patient had evaluable data at this timepoint | 0.9 (NA) — Only one patient had evaluable data at this timepoint

10. Secondary Outcome: Measurement of PK Parameter Terminal Half Life for MOv18 IgE
Description: Serum samples were analysed to determine the concentrations of MOv18 IgE using a previously developed ELISA method. Not all participants were analysed at all time points.
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | MOv18 IgE Cohort 1 | MOv18 IgE Cohort 2 | MOv18 IgE Cohort 3 | MOv18 IgE Cohort 4 | MOv18 IgE Cohort 5 | MOv18 IgE Cohort 6 | MOv18 IgE Cohort 7 Before Intra-Patient Dose Escalation | MOv18 IgE Cohort 7 After Intra-patient Dose Escalation
Number analyzed (Participants) | 2 | 5 | 5 | 2 | 2 | 1 | 1 | 1
Hour | NA (NA) — In one participant, MOv18 IgE could not be quantified in samples at any time point. In the other participant, MOv18 IgE could only be detected up to 7 hours postdose | 10.5 (0.6) | 9.9 (2.4) | 7.4 (0.3) | 9.2 (0.2) | 15.0 (NA) — Only one patient had evaluable data at this timepoint | 10.0 (NA) — Only one patient had evaluable data at this timepoint | NA (NA) — Half-life was not calculated for the 12 mg dose level due to a skewed value observed at the 6 h time point

11. Secondary Outcome: Measurement of the PK Parameter Mean Residence Time (MRT) of MOv18 IgE
Description: Serum samples were analysed to determine the MRT of MOv18 IgE following IV administration, using an ELISA method. Not all participants were analysed at all time points.
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | MOv18 IgE Cohort 1 | MOv18 IgE Cohort 2 | MOv18 IgE Cohort 3 | MOv18 IgE Cohort 4 | MOv18 IgE Cohort 5 | MOv18 IgE Cohort 6 | MOv18 IgE Cohort 7 Before Intra-Patient Dose Escalation | MOv18 IgE Cohort 7 After Intra-patient Dose Escalation
Number analyzed (Participants) | 2 | 5 | 5 | 2 | 2 | 1 | 1 | 1
Hour | NA (NA) — In one participant, MOv18 IgE could not be quantified in samples at any time point. In the other participant, MOv18 IgE could only be detected up to 7 hours postdose | 13.2 (1.1) | 12.5 (3.4) | 8.9 (0.3) | 11.4 (1.0) | 19.9 (NA) — Only one patient had evaluable data at this timepoint | 11.8 (NA) — Only one patient had evaluable data at this timepoint | NA (NA) — MRT was not calculated for the 12 mg dose level due to a skewed value observed at the 6 h time point

12. Secondary Outcome: Measurement of the PK Parameter Total Body Clearance (CLT) of MOv18 IgE
Description: Serum samples were analysed to determine the CLT of MOv18 IgE following IV administration, using an ELISA method. Not all participants were analysed at all time points.
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | MOv18 IgE Cohort 1 | MOv18 IgE Cohort 2 | MOv18 IgE Cohort 3 | MOv18 IgE Cohort 4 | MOv18 IgE Cohort 5 | MOv18 IgE Cohort 6 | MOv18 IgE Cohort 7 Before Intra-Patient Dose Escalation | MOv18 IgE Cohort 7 After Intra-patient Dose Escalation
Number analyzed (Participants) | 2 | 5 | 5 | 2 | 2 | 1 | 1 | 1
L/h | NA (NA) — In one participant, MOv18 IgE could not be quantified in samples at any time point. In the other participant, MOv18 IgE could only be detected up to 7 h postdose | 1.9 (0.8) | 1.6 (0.6) | 2.8 (0.5) | 1.7 (0.2) | 2.7 (NA) — Only one patient had evaluable data at this timepoint | 2.3 (NA) — Only one patient had evaluable data at this timepoint | 0.8 (NA) — Only one patient had evaluable data at this timepoint

13. Secondary Outcome: Measurement of the PK Parameter Volume of Distribution (Vss) of MOv18 IgE
Description: Serum samples were analysed to determine the Vss of MOv18 IgE following IV administration, using an ELISA method. Not all participants were analysed at all time points.
Time Frame: as for outcome 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: L
Arm/Group | MOv18 IgE Cohort 1 | MOv18 IgE Cohort 2 | MOv18 IgE Cohort 3 | MOv18 IgE Cohort 4 | MOv18 IgE Cohort 5 | MOv18 IgE Cohort 6 | MOv18 IgE Cohort 7 Before Intra-Patient Dose Escalation | MOv18 IgE Cohort 7 After Intra-patient Dose Escalation
Number analyzed (Participants) | 2 | 5 | 5 | 2 | 2 | 1 | 1 | 1
L | NA (NA) — In one participant, MOv18 IgE could not be quantified in samples at any time point. In the other participant, MOv18 IgE could only be detected up to 7 h postdose | 24.4 (10.2) | 18.7 (6.2) | 25.9 (5.4) | 20.1 (4.6) | 53.2 (NA) — Only one patient had evaluable data at this timepoint | 27.3 (NA) — Only one patient had evaluable data at this timepoint | 38.3 (NA) — Only one patient had evaluable data at this timepoint

ADVERSE EVENTS:
Time Frame: Safety data were collected from the date of written informed consent and continued until 70 days after the last dose of MOv18 IgE, an average (median) of 88.5 days (range: 13-181).
Arm/Group | MOv18 IgE Cohort 1 | MOv18 IgE Cohort 2 | MOv18 IgE Cohort 3 | MOv18 IgE Cohort 4 | MOv18 IgE Cohort 5 | MOv18 IgE Cohort 6 | MOv18 IgE Cohort 7
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/8 | 0/6 | 0/3 | 0/3 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 6/8 | 5/6 | 0/3 | 0/3 | 2/3 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 7/8 | 6/6 | 3/3 | 3/3 | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MOv18 IgE Cohort 1 (N=2) | MOv18 IgE Cohort 2 (N=8) | MOv18 IgE Cohort 3 (N=6) | MOv18 IgE Cohort 4 (N=3) | MOv18 IgE Cohort 5 (N=3) | MOv18 IgE Cohort 6 (N=3) | MOv18 IgE Cohort 7 (N=1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin test positive (Investigations) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MOv18 IgE Cohort 1 (N=2) | MOv18 IgE Cohort 2 (N=8) | MOv18 IgE Cohort 3 (N=6) | MOv18 IgE Cohort 4 (N=3) | MOv18 IgE Cohort 5 (N=3) | MOv18 IgE Cohort 6 (N=3) | MOv18 IgE Cohort 7 (N=1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (5)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 2 (3) | 2 (6) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 3 (3) | 2 (5) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (7) | 0 (0) | 2 (6) | 2 (9) | 3 (11) | 1 (4)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (10) | 0 (0) | 1 (6) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Secretion discharge (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 3 (8) | 3 (12) | 3 (12) | 3 (10) | 1 (3)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Xeroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/21/NCT02546921/Prot_000.pdf